CLINICAL TRIAL: NCT04447066
Title: Semicircular Canals Dysfunction Among Patients Hospitalized at the Rehabilitation Department
Brief Title: The Prevalence of Semicircular Canal Dysfunction Among Rehabilitation Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 255-20
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Vertigo; Dizziness
MeSH Terms: conditions — Vertigo; Dizziness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients hospitalized at the rehabilitation department
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention - VHIT will be used but without intervention

SUMMARY:
Patients hospitalized at the rehabilitation department at the hospital will fill a questionnaire regarding dizziness and ear diseases, and the Dizziness Handicap Inventory, and then will be examined by an ENT physician, followed by a video Head Impulse Test (vHIT) study.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old
* Hospitalized at the rehabilitation department

Exclusion Criteria:

* Blindness or loss of vision which is not corrected using glasses
* Past CVA with neurological remnants
* Movement disorder
* Lower body part weakness
* Limitation in neck movement
* Vestibular pathology diagnosed in the past 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized at the rehabilitation department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Video Head Impulse Test (vHIT) results | 1 year
  The results of the vHIT study in terms of gain and saccades

IPD SHARING:
Plan to Share IPD: No